CLINICAL TRIAL: NCT06385678
Title: A Phase IB/II Clinical Study on the Safety, Tolerability and Efficacy of HRS-4642 in Combination With Anti-tumor Medication in Subjects With Advanced Solid Tumors
Brief Title: A Study of HRS-4642 in Patients With Advanced Solid Tumors Harboring KRAS G12D Mutation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4642-201
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Advanced KRAS G12D Mutant Solid Tumors
MeSH Terms: interventions — Pemetrexed; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): For HRS-4642 in combination with Adebrelimab or in combination with Adebrelimab and chemotherapy for advanced solid tumors with KRAS G12D mutations.
  Interventions: Drug: HRS-4642; Drug: Adebrelimab; Drug: Pemetrexed Disodium for Injection、Cisplatin Injection、Carboplatin for Injection
- Arm 2 (Experimental): For HRS-4642 in combination with SHR-9839，for advanced solid tumors with KRAS G12D mutations.
  Interventions: Drug: HRS-4642; Drug: SHR-9839
- Arm 3 (Experimental): For HRS-4642 in combination with Cetuximab Solution for Infusion，for advanced solid tumors with KRAS G12D mutations
  Interventions: Drug: HRS-4642; Drug: Cetuximab Solution for Infusion

INTERVENTIONS:
Drug: HRS-4642 — administrated per dose level in which the patients are assigned
Drug: Adebrelimab — administrated per dose level in which the patients are assigned
  Arms: Arm 1
Drug: SHR-9839 — administrated per dose level in which the patients are assigned
  Arms: Arm 2
Drug: Pemetrexed Disodium for Injection、Cisplatin Injection、Carboplatin for Injection — administered as prescribed by the investigator.
  Arms: Arm 1
Drug: Cetuximab Solution for Infusion — administrated per dose level in which the patients are assigned
  Arms: Arm 3

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, and efficacy of HRS-4642 in combination with antitumor medicine in patients with advanced solid tumors harboring KRAS G12D mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. Male or female ≥ 18 years old and ≤75 years old.
3. ECOG performance status of 0-1.
4. With a life expectancy of ≥12 weeks.
5. With unresectable locally advanced or metastatic solid tumors harbouring with KRAS G12D mutation confirmed by central laboratory testing.
6. Need to provided tumor tissue samples for genetic testing.
7. Have at least one measurable lesion according to RECIST1.1, and the dose-escalation phase allows no measurable lesion.
8. Adequate laboratory parameters during the screening period.

Exclusion Criteria:

1. Accompanied by untreated or active central nervous system (CNS) metastases. Subjects with a history or current history of meningeal metastasis.
2. Systemic antitumor therapy was received 4 weeks before the start of the study.
3. Palliative radiotherapy was completed within 14 days before the first dose.
4. Toxicity and/or complications from previous interventions did not return to NCI-CTCAE level ≤1 or exclusion criteria.
5. Subjects with known or suspected interstitial pneumonia.
6. Moderate or severe ascites with clinical symptoms; Uncontrolled or moderate or higher pleural effusion or pericardial effusion.
7. Have poorly controlled or severe cardiovascular disease.
8. Subjects with active hepatitis B or active hepatitis C.
9. A history of immunodeficiency, including a positive HIV test, other acquired or congenital immunodeficiency disorders, or a history of organ transplantation.
10. The presence of uncontrolled mental illness and other conditions known to affect the completion of the study process, such as alcohol, drug or substance abuse, and criminal detention.
11. Any other factors that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate as judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Phase IB: Safety endpoints: adverse events (AEs). | 24 months
  Assess safety and tolerability by way of adverse events (CTCAE v5.0).
Phase IB： Maximum tolerated dose (MTD) | From Day 1 to Day 21
  Incidence and category of dose limiting toxicities (DLTs) during the first 21-day cycle of treatment.
Phase IB：Recommended phase 2 dose (RP2D) | 24 months
  RP2D will be determined on the basis of evaluation on safety, PK, efficacy data in dose escalation and dose expansion stages.
Phase II: Overall response rate (ORR). | 24 months.
  Evaluated by RECIST v1.1.

SECONDARY OUTCOMES:
Efficacy endpoints: Overall response rate (ORR). | 24 months
  Evaluated by RECIST v1.1.
Efficacy endpoints: Duration of response (DoR). | 24 months
  Evaluated by RECIST v1.1.
Efficacy endpoints: Disease control rate (DCR). | 24 months
  Evaluated by RECIST v1.1.
Efficacy endpoints: Progression free survival (PFS). | 24 months
  Evaluated by RECIST v1.1.
Efficacy endpoints: overall survival (OS). | 24 months
  Evaluated by RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided